CLINICAL TRIAL: NCT01526590
Title: A Pilot Study of the Effects of Contrast Enhanced Endoscopic Ultrasound on Determining Vascular Involvement in Pancreatic Lesions
Brief Title: Contrast Enhanced Endoscopic Ultrasound for Vascular Involvement in Pancreatic Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of support
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, James Hebert, Mackay-Page Professor of Surgery, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRMS_M11-203
Record Dates: First submitted 2012-01-10; First posted 2012-02-06 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Pancreatic Tumors
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Definity (Experimental): Patients enrolled in the study will undergo contrast enhanced endoscopic ultrasound of the pancreas with Definity contrast after they have undergone their standard of care endoscopic ultrasound of the pancreas.
  Interventions: Drug: Definity Contrast

INTERVENTIONS:
Drug: Definity Contrast — While the patient is still sedated from their EUS and before tissue sampling, the patient will receive a dose of Definity intravenously through their peripheral IV access after being agitated. The dose of Definity will be 10 microliters/kg given in one to two doses, and will not exceed 2cc.
  Other Names: Definity ultrasound contrast

SUMMARY:
In the US, pancreas cancer is the fifth leading cause of cancer related deaths. It was estimated to have taken 36,800 lives in 2010. Unfortunately, curing pancreatic cancer requires surgical removal. Surgical removal of the pancreas is associated with high morbidity and mortality, as well as high rates of complications. One way to aid surgeons in removing pancreatic tumors is by providing them with a good idea of where the tumor is located and what surrounding structures are involved. This currently happens through many different modalities of imaging; usually computed tomography (CT) and endoscopic ultrasound. Even with these forms of imaging (and sometimes others), surgeons will occasionally open a patient and find that the tumor cannot be removed due to its involvement with surrounding structures.

One way to avoid potentially unnecessary procedures or to help a surgeon navigate this delicate procedure would be to provide more detailed information about the tumor. Several of the techniques currently used to image the body have rapidly advanced over recent years. Typical advancements come through better resolution of the images or contrast to enhance desired parts of the images. Ultrasound has not seen such a two pronged advance. Ultrasound has seen substantial advances in resolution to enhance picture quality, but contrast has not been used clinically to assess pancreatic masses whereas it is for cardiologists to use contrast to look at potential defects in the heart.

The contrast that is used with ultrasound is different from that of CT scans. CT scanners use a dye that can be potentially hazardous. This dye can lead to serious kidney damage in some patients. Ultrasound contrast, on the other hand, is made of small micro bubbles filled with a harmless gas. Because of the way ultrasound works, these micro bubbles reflect the sound waves differently than the surrounding tissue and thus provide contrast between normal tissue and abnormal tissue. The contrast used in this study, Definity, and is the same contrast used by Cardiologists.

The CE-EUS will be used for research purposes only and will not be used for any clinical decision making. The surgeon will be blinded to the results of the research CE-EUS. The investigators will compare the research pre-operative contrast enhanced endoscopic ultrasounds images with already completed standard-of-care CT scans, the actual pancreatic involvement seen in surgery and the pathology reports.

DETAILED DESCRIPTION:
1. CT Scan of the abdomen - Standard Therapy

   a. The standard of care is that patients in question of pancreatic lesions undergo CT scanning. After a CT scan, if it appears that the pancreatic mass may be resectable, the standard protocol is to look at the pancreas while the patient is sedated with endoscopic ultrasound for diagnostic tissue sampling and further staging. For this reason, the endoscopist will not be blinded to the CT scan because it is the standard of care that they interpret the results of the EUS with that information.
2. Consent for Endoscopic Ultrasound (EUS) - Standard Therapy

   a. Before being sedated and having endoscopic ultrasound, all patients are informed about the risks of the procedure, alternatives, and what will be done. The patients who decide to undergo endoscopic ultrasound will sign a consent form. Our goal is to enroll 30 patients (This number is limited by both the amount of contrast received from Lantheus and the number of patients typically seen in a year. Ideally we will enroll as many as possible for the purposes of power).
3. Consent for Contrast Enhanced Endoscopic Ultrasound (CE-EUS) -- Performed exclusively for research purposes

   1. After the patient has been informed about the standard of care and signed a consent form, the patient will be asked if they wish to participate in an experimental study. If the patient is interested, they will be questioned about potential structural heart defects, congenital heart defects, recent worsening of heart or lung conditions, pulmonary hypertension, potential pregnancy, attempts to become pregnant, if they are nursing, or allergies to the contrast. If they report any of these relative contraindications, we will exclude them from participating in the study.
   2. If they are free of all of those relative contraindications, they will be provided information about the study (see included forms) and will be asked to sign a consent form as well as a HIPAA authorization.
4. EUS - Standard of Care

   1. At this point they will undergo an endoscopic ultrasound of the pancreas as per standard protocol. They will have a peripheral IV started by the endoscopic technician or nurse anesthetist. While the patient is being prepared, both research questionnaires (EUS and CE-EUS) will be filled out ahead of time with the exception of the findings, in order to reduce the time to complete the survey. The patient will be sedated in one of two ways. Either they will be consciously sedated with meperidine and midazolam under the surveillance of the attending gastroenterologist or they will have propofol based sedation under the surveillance of an anesthesiologist as per standard endoscopic ultrasound protocol.
   2. The patient will undergo their endoscopic ultrasound and video and images will be recorded.
5. EUS Questionnaire - Preformed exclusively for research purposes. Duration less than one minute.

   1. The endoscopist will then fill out a survey (see attached) to record their impressions of the tumor and the extent of its invasion into the vasculature. This should not take more than one minute. EUS criteria for vascular invasion will be loss of normal hyperechoic interface between the tumor and the vessel, irregular tumor and vessel interface, tumor within vessel lumen, vessel encasement, or collaterals with venous occlusion.
6. Decision about FNA - Standard of care, but important that it is done before CU-EUS a. If the endoscopist feels that FNA is warranted they will make the decision at this time.
7. CE-EUS - Experimental Procedure performed exclusively for research purposes

   a. Dosing of Contrast - procedure performed exclusively for research purposes i. While the patient is still sedated and before tissue sampling, the experimental aspect of the procedure will begin. At this time, they will receive a dose of Definity intravenously through their peripheral IV access after being agitated. The dose of Definity will be 10 microliters/kg given in one to two doses, and will not exceed 2cc. A saline flush will follow the injection of the contrast and a timer will be started. The remaining contrast will be properly disposed of in a sharps container.

   b. Recording of CE-EUS images - procedure performed exclusively for research purposes. Duration 3-4 minutes i. The endoscopist will perform an additional reading with the contrast and record a 3-4 minute segment for review later using the harmonic mode of the ultrasound probe at a mechanical index of 0.3. The mechanical index may need to be be optimized, however a previous study found 0.3 to be optimal. Aspects that will be analyzed later are sequence of filling (central vs peripheral), timing (arterial [0-30s], venous [60-180s], post-venous/equilibrium phase [>180s]), pattern of perfusion (homogenous vs heterogenous, and with or without defect) and degree of venous washout. After the experimental portion of the procedure the endoscopist will fill out a form (see attached) to record their impressions of the characteristics of the tumor with contrast. The images will be saved for further comparison with the CT scan and the pathology results at a later time.
8. FNA - Standard of care (if previously decided upon)

   a. If it was determined after the normal EUS but before the CE-EUS that the patient needed tissue sampling, the patient will then undergo the sampling in the standard fashion. If the patient was not to receive tissue sampling, the exam would be over. When the exam is finished the endoscopist will fill out the remaining questionnaire while the patient recovers.
9. Patient recovery in Endoscopy Suite - Standard of Care
10. Patient transport to recovery room - Standard of Care

    1. After the patient recovers in the endoscopy room, the patient will be transported to the recovery room where they will be monitored for at least 30 minutes. The patient will be informed of the findings of their EUS per standard care. The patient will not be informed of the findings of CE-EUS as the significance is unknown.
    2. If an incidental lesion is found on EUS then the patient will undergo the appropriate follow-up for that lesion as per standard protocol. If an incidental finding is not apparent on EUS or CT, but happens to show up with the CU-EUS, the patient will be informed of the finding and its unknown significance.
11. Radiologist's Interpretation - Research purposes only

    a. After CE-EUS and EUS, the images will be randomly ordered and interpreted by a radiologist. An excel sheet will be made and the studies will be placed into three separate blocks in chronological order Participant 1-10, 11-20, and 21-30. In a separate column a random number generator will order the first block of 1-10's EUS into a random order for and then again a different random order for CE-EUS. The radiologist will fill out the attached questionnaire. The Surgeon will be blinded to these readings as they are for research purposes only and not the standard of care.
12. Surgery - Standard of Care with questionnaire after the procedure for research purposes

    a. The surgeon will record their impressions of the vascular involvement of the tumor on the attached questionnaire after the surgery.
13. Pathology review - Standard of care a. If the patient has pathology sent from surgery, the surgeon will label the vessels encompassed and the pathologist will report whether there was invasion into the vasculature. We will retrospectively review the pathology results of the surgery for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pancreatic lesion undergoing EUS for diagnosis and pre-operative assessment.

Exclusion Criteria:

* Pregnant women, breastfeeding women and individuals with metastatic lesions on CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Lesion Margin | Up to six months

SECONDARY OUTCOMES:
Sequence of filling | Up to six months
Pattern of Perfusion | Up to six months
Degree of venous washout | Up to six months

CONTACTS AND LOCATIONS:
Overall Officials: James Hebert, M.D., Principal Investigator — University of Vermont/Fletcher Allen Healthcare
Locations (1):
- Fletcher Allen Healthcare, Burlington, Vermont, United States